CLINICAL TRIAL: NCT05468411
Title: Effects of Oral Application of Miracle Fruit Pill Before Eating Food on Food Likings and Energy Intake in Diabetic or Prediabetic Patients: A Randomized Crossover Trial
Brief Title: Effects of Miracle Fruit Pill Application on Food Likings and Energy Intake in Diabetic or Prediabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queens College, The City University of New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: PSC-CUNY 62192-00-50
Record Dates: First submitted 2022-07-06; First posted 2022-07-21 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Diabetes; PreDiabetes
Keywords: Miracle fruit; Alternative sweetener; Taste liking; Energy intake; Placebo
MeSH Terms: conditions — Diabetes Mellitus; Prediabetic State

STUDY DESIGN:
Intervention Model Description: This study is a randomized crossover trial that has two interventions (miracle fruit pill and placebo). This means that participants have a 100% chance of getting both applications.
  Participants are asked to participate in a total of six sessions (Part 1: session 1, 2, & 3, Part 2: session 4, 5, & 6). Participants are randomly assigned to either of two interventions (miracle fruit and placebo) in part 1 and their assignment are switched from one application to another in part 2.
Who Masked: Participant
Masking Description: The taste modifying function of miracle fruit as a sweetness enhancer is masked. Participants are told that they are participating in a study developing a dietary supplement for diabetic patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Miracle fruit pill (Active Comparator): A freeze-dried miracle fruit pill is orally administered prior to eating food samples.
  Interventions: Other: Oral application of miracle fruit pill; Other: Oral application of sugar candy
- Sugar candy (Placebo Comparator): A chewable sugar candy is orally administered as a placebo prior to eating food samples.
  Interventions: Other: Oral application of miracle fruit pill; Other: Oral application of sugar candy

INTERVENTIONS:
Other: Oral application of miracle fruit pill — Miracle fruit has a taste modifying function from sourness to sweetness when it is exposed to an acidic environment. To activate the miracle fruit's function, a miracle fruit pill should be orally administered to coat taste buds prior to eating sour food. Thus, participants are instructed to place a miracle fruit pill is on their tongue, and roll the pill around their mouth to allow full contact of the pill with the surface of the oral cavity without chewing until the pill completely dissolved. A miracle fruit pill is administered prior to eating.
Other: Oral application of sugar candy — To simulate the miracle fruit's function as a placebo, a chewable sugar candy that has a similar appearance to miracle fruit pill is orally administered. The same protocol that is used in miracle fruit intervention is followed in this placebo intervention but with a chewable sugar candy. Participants are instructed to place a sugar candy is on their tongue, and roll the candy around their mouth to allow full contact of the candy with the surface of the oral cavity without chewing until the candy completely dissolved. A sugar candy is administered prior to eating.

SUMMARY:
The high prevalence of diabetes and prediabetes has increased the demand for nonnutritive sweeteners in recent years. Miracle fruit has been considered a healthy alternative sweetener for diabetic patients due to its sweetness-enhancing effects and high antioxidant activity. The purposes of this study are to examine whether the miracle fruit pill application to mouth prior to food consumption could improve the likings of different types of sour food (green apple, goat cheese, lemonade, cucumber pickle, and plain fat-free yogurt) and meals (breakfast, lunch, and dinner), and reduce energy intakes at the meals. Fifty volunteers (25 men and 25 women) aged 45 to 75 years with diabetes or prediabetes participate in the study. In this study, two interventions (miracle fruit and placebo) are provided, and all participants receive both applications. Participants are randomly assigned to one of the two interventions in part 1 and the assignment is switched from one application to another in part 2. The study hypotheses of this study are that the miracle fruit intervention improves the likings for sour foods and meals more than the placebo does; The miracle fruit intervention also reduces energy intakes from the meals more than the placebo does. Participants are asked to participate in a total of 6 sessions (1 hour/session, 1 session/day, Part 1: session 1, 2, & 3, Part 2: session 4, 5, & 6). Each session consists of two 30-min assessments, which are liking tests and meal intake assessment. The potential participants who have known food allergies or food intolerances are screened through consented screening procedure. If unknown food allergies or intolerances unintentionally become present during the study, medical help will be sought immediately. Participants may enjoy food samples and meals provided in this study and benefit by learning more about their acceptances for miracle fruit pill as an alternative sweetener. The results of this research are expected to develop generalizable knowledge about the miracle fruit's potential to improve the food palatability for people with diabetes or prediabetes.

DETAILED DESCRIPTION:
Due to the rise in rates of obesity and diabetes in recent years, the consumer demand for alternative sweetener is growing especially among people with diabetes or prediabetes. Given the need for alternative sweeteners, miracle fruit (Synsepalum dulcificum) may be a good candidate to fulfill the demand. Miracle fruit has been used as a sweet enhancer for thousands of years by the natives in Western Africa without any reports of adverse effects. The red, cranberry-sized miracle fruit is named for its unique ability to transform sour taste into sweet. In addition to the miracle fruit's taste modification function, miracle fruit has valuable antioxidant activities that can be applied for functional food and has also been studied to improve insulin resistance induced by fructose-rich chow in rats. With the potential health benefit of miracle fruit, miracle fruit has been considered as a healthy alternative sweetener that can meet diabetic patients' needs. However, for the practical applications of miracle fruit for diabetic diet, the acceptability of miracle fruit and its effect on energy intake need to be examined among diabetic patients. Fresh miracle fruits are highly perishable, and they cannot be cooked because the taste modifying effect found in the pulp of the miracle fruit is due to a protein, which is deactivated by heat. For these reasons, a freeze-dried pill form of miracle fruit needs to be applied on a tongue to coat taste buds before food is consumed. Therefore, in this study, the effects of oral application of miracle fruit pill are compared with placebo (sugar candy) on the likings of different sour food products (green apple, goat cheese, lemonade, cucumber pickle, and plain fat-free yogurt) and meals (breakfast, lunch, and dinner), and energy intakes from the meals in people with diabetes or prediabetes. A total of 50 patients aged 45 to 75 years who have been diagnosed with diabetes or prediabetes (25 men and 25 women) participate in this study. They should be nonsmokers; not have food allergies or food intolerances; not be diagnosed with taste disorders; not be pregnant; not breastfeed; and not use medications that could affect taste perception and food intake. This study is a randomized placebo-controlled crossover trial. As an intervention, a miracle fruit pill is orally administered prior to eating food samples. The same protocol is followed in the control group but with placebo (sugar candy). Participants are asked to participate in a total of six 1-hour sessions (1 session/day). Participants are randomly assigned to either of two applications (miracle fruit and placebo) in part 1 and one week after part 1 (1-week washout), their intervention assignment is switched from one application to another in part 2. Each part/intervention consists of 3 sessions and each session consists of two assessments (liking tests and meal intake assessment). In each part/intervention, each participant performs the liking tests for five sour foods in triplicate and consumes breakfast, lunch, and dinner meals once. The order of the experiments in each session is as follows: 1. preliking test; 2. miracle fruit pill/placebo administration; 3. postliking test; and 4. meal intake. At the liking tests, the pre- and postlikings of overall, flavor, texture, and aftertaste for all 5 sour food samples are assessed using a 9-point hedonic scale (1=dislike extremely, 9=like extremely). For the meal intake assessment, standardized breakfast, lunch, and dinner meals are provided to participants according to the experimental design. During the meal intake session, participants are allowed to consume any food, beverage, or condiments, including sweeteners that are provided at the session. All foods and beverages that are consumed by each participant at the meals are weighed, and the energy intakes from the meals are calculated using the food weight via online nutrient tracker.

ELIGIBILITY:
Inclusion Criteria:

* Having a score of 5 or higher on the 'Prediabetes Risk Test' provided by the American Diabetes Association and the Centers for Disease Control and Prevention
* Having been diagnosed with prediabetes or diabetes by doctor

Exclusion Criteria:

* Smoking
* Having food allergies or food intolerances
* Being diagnosed with taste disorders
* Being pregnant
* Breastfeeding
* Using medications that could affect taste perception and food intake

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in food liking from pre- to post-intervention | The pre-liking test (10 minutes),intervention application & break (10 minutes), and post-liking test (10 minutes) are conducted consecutively and completed within a session.
  Changes in food liking for sour food samples (green apple, goat cheese, lemonade, cucumber pickle, and plain fat-free yogurt) are measured by comparing pre-and post-liking scores for sour food samples. Before the intervention (oral application of miracle fruit pill or placebo sugar candy) is applied, the pre-liking is assessed by tasting each food sample. After the pre-liking test is done, the intervention is applied. It takes approximately 5 minutes for intervention pills (miracle fruit pill or sugar candy) to dissolve. After the oral application/intervention is completed, the post-liking is assessed in the same way as the pre-liking. The pre- and post-likings for overall, flavor, texture, and aftertaste are evaluated using a 9-point hedonic scale (1=dislike extremely, 9=like extremely). For "aftertaste pleasantness", the 'no aftertaste detected' answer option is additionally provided.
Energy intake from meals | Each participant's food intake is measured for 30 minutes.
  All foods and beverages that are served to each participant at the meal sessions are preweighed, and food intake is assessed by measuring their remaining food and beverages. The energy intake of each participant is calculated using the food weight on an online nutrient analysis site.
Overall liking for meals | Immediately after the energy intake measurement is done, overall liking for each meal is evaluated.
  Overall liking for each of meals (breakfast, lunch, and dinner) is evaluated using a 9-point hedonic scale (1=dislike extremely, 9=like extremely).

CONTACTS AND LOCATIONS:
Overall Officials: Sungeun Choi, PhD, Principal Investigator — Queens College, CUNY
Locations (1):
- Korean Community Services of Metropolitan New York, Inc., Bayside, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD in a publication.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 6 months after article publication and the data will be available for up to 12 months
Access Criteria: Data obtained through this study may be provided to qualified researchers engaging in independent scientific research. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party. For more information or to submit a request, please contact Dr. Sungeun choi (sungeun.choi@qc.cuny.edu).

REFERENCES:
- [Derived] Choi S, Park T. Feasibility and acceptability of miracle fruit application prior to the consumption of sour-tasting foods as a weight-loss strategy in adults with diabetes or prediabetes: A randomized crossover trial. Appetite. 2023 Dec 1;191:107046. doi: 10.1016/j.appet.2023.107046. Epub 2023 Sep 17. PMID 37726068